CLINICAL TRIAL: NCT00369980
Title: Diagnostic Usefulness of Fluorine-18-α-Methyltyrosine PET in Combination With 18F-FDG in Sarcoidosis Patient
Status: Completed | Type: Observational
Sponsor: Gunma University (Other)
Other Study IDs: GunmaU
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
L-[3-18F]-α-methyltyrosine (FMT) is amino-acid tracer for positron emission tomography (PET), and is used for tumor detection because malignant tumor cells accumulate 18F-FMT based on the increased expression of amino-acid transporter. This study was conducted to investigate a usefulness of 18F-FMT PET in combination with 18F-FDG PET for the diagnosis of sarcoidosis in patients with suspected malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were required to have histologically proven noncaseating epithelioid cell granuloma and at least one disease that the possibility of coexistent malignancy could not be excluded as follows; 1) extrapulmonary lesions mimicking malignant diseases including systemic lymphadenopathy, hepatosplenic involvement, or other lesions, 2) multiple nodular lesions mimicking pulmonary metastasis, 3) the occurrence of BHL in cancer patient.

Exclusion Criteria:

* The patients that PET imaging using 18F-FDG and 18F-FMT was performed before establishment of the final diagnosis of sarcoidosis, patients undergoing treatment for sarcoidosis before the PET study, and patient having diabetes mellitus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: kyoichi kaira, MD, Principal Investigator — Gunma University Graduate School of Medicine
Locations (1):
- Gunma University Graduate School of Medicine, Gunma, Japan

REFERENCES:
- [Derived] Kaira K, Oriuchi N, Otani Y, Yanagitani N, Sunaga N, Hisada T, Ishizuka T, Endo K, Mori M. Diagnostic usefulness of fluorine-18-alpha-methyltyrosine positron emission tomography in combination with 18F-fluorodeoxyglucose in sarcoidosis patients. Chest. 2007 Apr;131(4):1019-27. doi: 10.1378/chest.06-2160. PMID 17426205